CLINICAL TRIAL: NCT03417622
Title: Surgical Resection Margin According to the Post-treatment Tumor Volume Versus the Pre-treatment Tumor Volume in Breast Conservative Surgery for Invasive Breast Cancer Patients Receiving Primary Systemic Therapy: Randomized Controlled Trial
Brief Title: Wide Margin vs. Narrow Margin in Postneoadjuvant Lumpectomy
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Principal Investigator, Osama Hussein, Professor of surgery (surgical oncology), Mansoura University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R.18.02.33
Record Dates: First submitted 2018-01-24; First posted 2018-01-31 (Actual); Last update posted 2021-02-25 (Actual); Status verified 2021-02

CONDITIONS: Breast Cancer
Keywords: resection margin; neoadjuvant therapy; breast conservative surgery; locally advanced breast cancer
MeSH Terms: conditions — Breast Neoplasms; Margins of Excision | interventions — Neoadjuvant Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Post-treatment volume-resection margin (Experimental): Lumpectomy is performed with resection margin of the clinically / radiologically identifiable post-treatment tumor.
  Interventions: Procedure: Bracketing; Drug: Neoadjuvant therapy; Procedure: Post-treatment volume margin resection
- Pre-treatment volume-resection margin (Active Comparator): Lumpectomy is performed with resection margin of the bracketed tissue.
  Interventions: Procedure: Bracketing; Drug: Neoadjuvant therapy; Procedure: Pre-treatment volume margin resection

INTERVENTIONS:
Procedure: Bracketing — At the beginning of therapy, ultrasonographic examination is used to measure the tumor in three dimensions and bracket the tumor using 4-6 metal clips which will serve as markers for the initial tumor extent in case of tumor shrinkage in response to systemic treatment.
Drug: Neoadjuvant therapy — All patients will receive primary systemic therapy according to the current institutional guidelines. Drugs include cytotoxic chemotherapy, hormonal therapy and/or anti-HER2/neu therapy as indicated.
Procedure: Post-treatment volume margin resection — The lumpectomy resection margin is planned according to the identifiable tumor at operation. The initial extent of the tumor at diagnosis is not taken in account. If there is complete clinical response to systemic therapy (i.e. no identifiable tumor), the center of the bracketed tissue is biopsied.
  Arms: Post-treatment volume-resection margin
Procedure: Pre-treatment volume margin resection — The lumpectomy includes the whole bracketed tissue to take in account the initial tumor extent before systemic therapy.
  Arms: Pre-treatment volume-resection margin

SUMMARY:
Breast cancer patients often receive systemic drugs as the initial curative treatment of their disease. The initial systemic therapy leads to a variable degree of tumor shrinkage. At present, there is no evidence-based consensus among breast surgeons on the optimal extent of resection after considerable tumor shrinkage and whether resection margin should be designed according to the tumor extent before treatment or the extent after treatment. This trial will help determine the optimal extent of resection in tumors that exhibits a significant change in volume after primary systemic therapy.

DETAILED DESCRIPTION:
Primary systemic (neoadjuvant) therapy (NAT) is a widely practised curative treatment for invasive breast cancer. Neoadjuvant chemotherapy (before surgery) and adjuvant chemotherapy (after surgery) had equivalent survival rates in major randomized trials. In these studies, preoperative systemic therapy increased the patient's chance to achieve breast conservation. The down side was a clear trend towards increased ipsilateral breast tumor recurrence. Preoperative chemotherapy leads to patchy, irregular cell death known as honeycomb effect and thus may lead to a misleading false negative resection margin of a tumorectomy operation. Even with the advent of oncoplastic techniques which allowed larger resection volumes with satisfactory cosmetic results, rates of re-excision, mastectomy and local relapse did not differ from those after traditional lumpectomy operations. As of today, there is no consensus -based on evidence- on the optimal width of margin in patients who are offered breast conservative surgery (BCS) after systemic therapy. In view of the current uncertainty and lack of evidence, The present trial is designed to answer the following question (Specific aim): Does planning the resection margin according to the pre-treatment tumor extent improve the local recurrence rate in patients receiving breast conservative surgery after systemic therapy?

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven diagnosis of invasive adenocarcinoma of the breast.
* Tumor stage T 1-4b
* Nodal stage N 0-2
* ASA (American Society of Anesthesiologists) class I-II

Exclusion Criteria:

* Patients opting for mastectomy.
* Patients advised for mastectomy by the treating physician.
* Patients opting for primary surgical treatment.
* Patients advised for primary surgical treatment by the treating physician.
* Metastatic patients.
* Multifocal tumors.
* Lobular neoplasia.
* Current pregnancy or pregnancy less than 6 months from the enrollment date.
* Active second cancer.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 370 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2026-08-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Local recurrence rate. | at 60 months after the date of diagnosis.
  The rate of local recurrence at five years.

SECONDARY OUTCOMES:
Local disease-free survival. | up to 60 months from the date of diagnosis.
  The proportion of patients who remain free of local disease recurrence.
Disease-free survival. | up to 60 months from the date of diagnosis.
  The proportion of patients who remain free of disease recurrence.
Overall survival. | up to 60 months from the date of diagnosis.
  The proportion of patients who are alive.

OTHER OUTCOMES:
Mastectomy rate. | at 6 months from the date of first surgical intervention.
  The proportion of patients who undergo mastectomy after failed conservative surgery.
Cosmetic score. | at 6 months from the date of first surgical intervention.
  Numeric score description of the cosmetic outcome of breast conservative surgery.

CONTACTS AND LOCATIONS:
Locations (1):
- Mansoura University Oncology Center, Al Mansurah, DK, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Zhou X, Li Y. Local Recurrence after Breast-Conserving Surgery and Mastectomy Following Neoadjuvant Chemotherapy for Locally Advanced Breast Cancer - a Meta-Analysis. Breast Care (Basel). 2016 Oct;11(5):345-351. doi: 10.1159/000450626. Epub 2016 Oct 14. PMID 27920628
- [Background] Gnant M, Harbeck N, Thomssen C. St. Gallen/Vienna 2017: A Brief Summary of the Consensus Discussion about Escalation and De-Escalation of Primary Breast Cancer Treatment. Breast Care (Basel). 2017 May;12(2):102-107. doi: 10.1159/000475698. Epub 2017 Apr 26. PMID 28559767